CLINICAL TRIAL: NCT04023266
Title: A Pilot Randomized Controlled Trial of Intravenous N-acetyl Cysteine in Patients Undergoing Pharmaco-invasive Reperfusion Early After an ST-segment Elevation Myocardial Infarction
Brief Title: A Pilot Randomized Controlled Trial of Intravenous N-acetyl Cysteine in STEMI
Acronym: PANACEA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00087545
Record Dates: First submitted 2019-07-09; First posted 2019-07-17 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-07

CONDITIONS: STEMI
Keywords: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Drugs, Generic

STUDY DESIGN:
Intervention Model Description: Investigator-initiated prospective, single-center, double- arm non-blinded randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: The clinical outcomes assessor reading the cardiac MRI would be blinded to the study arm allotment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous N-Acetylcysteine arm (Experimental): On arrival at the recruiting hospital, eligible and consenting STEMI patients randomly allocated to the experimental arm would be administered an intravenous N-Acetylcysteine bolus of 1200 mg over 0.5 hours (in 5% Dextrose) followed by 600mg/hour for the remaining 47.5 hours (in 5% dextrose). A total N-acetylcysteine dose of 29.7 grams is administered over 48 hours.
  Interventions: Drug: Intravenous N-Acetylcysteine
- Control arm (No Intervention): Patients randomized to this arm would receive no experimental therapies and would continue to receive all standard guideline recommended medical therapies and interventions.

INTERVENTIONS:
Drug: Intravenous N-Acetylcysteine — Intravenous N-acetyl cysteine bolus and infusion as described in the experimental arm.
  Other Names: Generic
  Arms: Intravenous N-Acetylcysteine arm

SUMMARY:
The PANACEA trial is an investigator-initiated prospective, single-center, two-arm, non-blinded pilot randomized controlled trial of high-dose IV N-Acetylcysteine therapy used as an adjunct to pharmaco-invasive reperfusion in patients presenting early after a large STEMI.

DETAILED DESCRIPTION:
Patients presenting with ST-segment elevation myocardial infarction within 3 hours of symptom onset and satisfying all of the inclusion criteria after informed consent would be randomly allocated to either intravenous N-Acetylcysteine or standard treatment using a 1:1 allocation ratio. Those randomized to IV N-Acetylcysteine would be administered a bolus of 1200 mg over 0.5 hours (in 5% Dextrose) followed by 600mg/hour for the remaining 47.5 hours (in 5% dextrose). A total N-acetylcysteine dose of 29.7 grams is administered over 48 hours. The infusion is continued during the primary percutaneous coronary intervention. Patients would be followed up for a minimum of 90 days. The primary clinical endpoint will be myocardial infarct size measured by late gadolinium enhancement CMR imaging at 3-5 days from first medical contact. Primary feasibility outcome will be the rate of recruitment, the number of patients undergoing cardiac MRI within the stipulated time frame, and completeness of the study data collection.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting with STEMI within 3 hours of symptom onset and satisfying all of the following criteria:

1. Patient age ≥ 18 years
2. Have received thrombolysis, with intend to pursue a pharmaco-invasive reperfusion strategy. Onset of chest pain to reperfusion time of < 3hrs.
3. STEMI involving anterior and/or inferior wall
4. An absence of baseline Q-waves on the initial ECG: The presence of Q waves defined at baseline using the Selvester QRS screening criteria
5. Have a high-risk STEMI ECG defined as:

   * ≥2mm ST-segment elevation in 2 anterior or lateral leads; or
   * ≥2 mm ST-segment elevation in 2 inferior leads coupled with ST-segment depression in 2 contiguous anterior leads for a total ST-segment deviation of ≥4 mm

Exclusion Criteria:

1. Previous myocardial infarction
2. Known to have moderate to severe LV systolic dysfunction (LV EF< 45%)
3. Known allergy to thrombolytic therapy or NAC
4. Presence of left bundle branch block
5. Cardiogenic shock (defined as systolic blood pressure of < 90mm Hg, for at least 30 minutes, not responsive to fluid resuscitation)
6. Permanent pacemaker or cardioverter defibrillator implanted previously
7. Patients with contra-indications to thrombolytic therapy
8. Patients with loss of consciousness or confusion
9. Patients with known chronic kidney disease (GFR < 30ml/min/m2) or on dialysis
10. Current pregnancy
11. Planned therapy with primary PCI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Myocardial infarct size | 3-5 days after first medical contact
  The primary clinical endpoint will be myocardial infarct size measured by late gadolinium enhancement CMR imaging at 3-5 days from first medical contact.
Feasibility outcomes | Assessed at the end of the study
  Primary feasibility outcomes would include the rate of recruitment, the number of patients undergoing cardiac MRI within the stipulated time frame, and completeness of the study data collection.

SECONDARY OUTCOMES:
Myocardial salvage | 3-5 days after infarction
  Myocardial salvage as measured by T2-weighted short tau inversion recovery on CMR assessed at 3-5 days after infarction
Left ventricular ejection fraction | 3-5 days after infarction
  Left ventricular ejection fraction on CMR at 3-5 days
ST-segment elevation resolution | 90-minutes after thrombolysis
  ST-segment elevation resolution at 90 minutes after thrombolysis as assessed by the worst lead on electrocardiogram (ECG core lab).
TIMI frame count in infarct related artery | During index coronary angiogram which will be performed within 24 hours of admission
  TIMI frame count on baseline coronary angiogram in the infarct-related artery
Creatine kinase MB area under the curve | 24 hours after admission
  Creatine kinase MB area under the curve through 24 hours
Von Willebrand factor fragmentation | At the time of angiography, assessed up to 7 days from admission
  The proportion of Von Willebrand factor multimers in the low, intermediate and high molecular weight form at the time of angiography
Bleeding | From time of randomization until the date of discharge or date of death from any cause, whichever came first, assessed up to 90 days
  Bleeding research consortium type II, III and V bleeding; safety outcome
Allergic reactions | From time of randomization, upto 48 hours
  Allergic reactions including hypotension (SBP< 90 mm Hg or a fall in BP >30 mm Hg below baseline), urticaria, flushing, wheezing and/or angioedema

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Graham, MD. FRCPC, Study Chair — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data regarding IPD will be made available on reasonable request
Supporting Information: Study Protocol, ICF
Time Frame: ON publication of trial the study protocol will be detailed. The ICF has been uploaded on this site.
Access Criteria: Study protocol will be published

DOCUMENTS (1):
  • Informed Consent Form (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT04023266/ICF_000.pdf